CLINICAL TRIAL: NCT00106951
Title: Effects of Neighborhood SES on Coronary Heart Disease Burden in Communities - Ancillary to ARIC
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kathryn Rose, Adjunct Associate Professor, University of North Carolina, Chapel Hill
Other Study IDs: 1292; R01HL080287 (NIH)
Record Dates: First submitted 2005-04-01; First posted 2005-04-04 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
Keywords: Surveillance; coronary heart disease; neighborhood SES
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the role of racial and socioeconomic disparities in coronary heart disease (CHD) mortality in the United States.

DETAILED DESCRIPTION:
BACKGROUND:

Despite strong decreases in coronary heart disease (CHD) mortality over past decades, there is evidence that racial and socioeconomic disparities in CHD mortality are increasing. CHD surveillance efforts that examine trends within these population subgroups are an important first step in quantifying and reducing disparities. The Atherosclerosis Risk in Communities (ARIC) Study has monitored rates and trends in validated hospitalized myocardial infarction and fatal CHD among black and white adults aged 35 to 74 years in four U.S. communities since 1989.

DESIGN NARRATIVE:

The study will expand the scope of ARIC surveillance by examining variations in the rates and temporal trends in CHD by socioeconomic status (SES), measured at the level of census tract. For CHD events already included in ARIC surveillance (1992-2002), addresses will be obtained from medical records and death certificates and geocoded so that they can be matched with identifiers for census based geographical areas. The ARIC study will contribute yearly updates of abstracted CHD events and addresses for subsequent years (2003-2005). Each event will be linked with census tract level SES indicators available from the 1990 and 2000 censuses. This novel effort will permit an examination of disparities by SES in rates and trends in fatal CHD, hospitalized myocardial infarction, case fatality, use of invasive cardiac procedures and prescription of efficacious medication at time of hospital discharge. In addition, the extent to which racial disparities in CHD and associated treatments are explained by SES will also be explored.

ELIGIBILITY:
hospitalized and fatal coronary heart disease cases eligibility: within 4 defined geographic areas and ages 35 to 74 years of age

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community surveillance of adults in four communities in the US
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2005-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Rose, PhD, Principal Investigator — UNC (Adjunct)

REFERENCES:
- [Result] Foraker RE, Rose KM, Kucharska-Newton AM, Ni H, Suchindran CM, Whitsel EA. Variation in rates of fatal coronary heart disease by neighborhood socioeconomic status: the atherosclerosis risk in communities surveillance (1992-2002). Ann Epidemiol. 2011 Aug;21(8):580-8. doi: 10.1016/j.annepidem.2011.03.004. Epub 2011 Apr 23. PMID 21524592
- [Result] Foraker RE, Rose KM, Whitsel EA, Suchindran CM, Wood JL, Rosamond WD. Neighborhood socioeconomic status, Medicaid coverage and medical management of myocardial infarction: atherosclerosis risk in communities (ARIC) community surveillance. BMC Public Health. 2010 Oct 21;10:632. doi: 10.1186/1471-2458-10-632. PMID 20964853
- [Result] Rose KM, Suchindran CM, Foraker RE, Whitsel EA, Rosamond WD, Heiss G, Wood JL. Neighborhood disparities in incident hospitalized myocardial infarction in four U.S. communities: the ARIC surveillance study. Ann Epidemiol. 2009 Dec;19(12):867-74. doi: 10.1016/j.annepidem.2009.07.092. Epub 2009 Oct 7. PMID 19815428
- [Result] Foraker RE, Rose KM, McGinn AP, Suchindran CM, Goff DC Jr, Whitsel EA, Wood JL, Rosamond WD. Neighborhood income, health insurance, and prehospital delay for myocardial infarction: the atherosclerosis risk in communities study. Arch Intern Med. 2008 Sep 22;168(17):1874-9. doi: 10.1001/archinte.168.17.1874. PMID 18809814